CLINICAL TRIAL: NCT06452927
Title: Endoscopic Enucleation of the Prostate in Patients With Urodynamically Proven Detrusor Underactivity/Acontractility
Brief Title: EEP in Patients With Urodynamically Proven DU/DA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EEPiDuDa Study Group (Network)
Responsible Party: Principal Investigator, Pawel Trotsenko, Dr. med. Dr. med. univ., EEPiDuDa Study Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EEPiDuDa 1.0 - 2024
Record Dates: First submitted 2024-05-23; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Lower Urinary Tract Symptoms; Lower Urinary Tract Obstructive Syndrome; Detrusor Underactivity; Detrusor Areflexia; Prostatic Hyperplasia
Keywords: Endoscopic Enucleation of the Prostate; BipoEP; ThuLEP; Detrusor Underactivity; Detrusor Acontractility; HoLEP; Urodynamics; Pressure Flow Study
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Underactive; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic Enucleation of the Prostate (Other): Patients with urodynamically proven Detrusor Underactivity/Acontractility, who undergo endoscopic enucleation of the prostate (EEP).
  Interventions: Procedure: Endoscopic enucleation of the prostate

INTERVENTIONS:
Procedure: Endoscopic enucleation of the prostate — Endoscopic enucleation of the prostate, regardless of energy source.
  Also see:
  * Enucleation is enucleation is enucleation is enucleation
  * PMID: 27585786 DOI: 10.1007/s00345-016-1922-3

SUMMARY:
The aim of this project is to create und evaluate a multicentral, retro-/prospective database for patients with urodynamically proven detrusor underactivity (DU) or acontractility (DA) secondary to a non-neurogenic aetiology, who undergo endoscopic, anatomic enucleation of the prostate (EEP).

DETAILED DESCRIPTION:
Background:

As one of the most common urological diseases benign prostatic hyperplasia (BPH) affects about ¾ of men in the seventh decade and is associated with major impact on quality of life (QoL) of patients as well as with substantial costs for the health care. For many patients suffering from lower urinary tract symptoms (LUTS) medical therapy, such as the use of α1-blockers, is initially successful, but surgical therapy becomes necessary when medical therapy fails and results / function remain unsatisfactory. Dependent on prostate volume (PV), different surgical techniques are available for treatment. For substantially enlarged glands open prostatectomy (OP) dominated as the oldest surgical procedure for many years. However, OP is associated with significant complications, and is currently recommended by the European Association of Urology (EAU) only in the absence of laser-assisted endoscopic enucleation options.

Among these patients, the presence of detrusor underactivity (DU) and detrusor acontractility (DA) represents a particularly challenging condition since no medical treatment is available. Due to this, efforts were focused on maximal surgical reduction of bladder outlet resistance to ensure efficient bladder emptying. The limited data on this topic showed promising outcomes for patients receiving holmium laser enucleation of the prostate (HoLEP). Therefore, the aim of this project is to evaluate the efficacy of EEP as a surgical approach for patients with DU/DA, regardless of PV or enucleation device/method.

Projekt objectives:

* Creating a multicentral, retro-/prospective database for patients with urodynamically proven detrusor underactivity (DU) or acontractility (DA) secondary to a non-neurogenic aetiology, who undergo EEP.

  * Phase 1: retrospective (patients with urodynamically proven, meeting inclusion criteria, and postoperative outcome according to material and methods from existing patient chart.
  * Phase 2: prospective capture of patient's data according to material and methods.
* Estimated cohort-size: based on available data set.
* Powering of phase 2 based on the retrospective cohort.
* Evaluating EEP as a surgical approach for patients with DU/DA, regardless of PV or energy source for endoscopic EEP.
* Enhancing importance of preoperative urodynamics as a tool for precision medicine in LUTS

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic enucleation of the prostate in patients with DU/DA secondary to a non-neurogenic aetiology:

  * Detrusor underactivity (DU) defined urodynamically as a bladder contractility index (BCI) of <100.
  * Detrusor acontractility (DA) defined urodynamically as the absence of a detrusor contraction despite filling to bladder capacity.

Exclusion Criteria:

* Neurogenic aetiology for DU/DA (Parkinson, stroke…)
* Other surgical approaches for the treatment of benign prostate hyperplasia (Aquaablation, open enucleation of the prostate, open prostatectomy, transurethral resection of the prostate...)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Residual volume | 2 months after surgery
  Determined by sonography (ml)
Residual volume | 1 year after surgery
  Determined by sonography (ml)
International Prostate Symptom Score (IPSS) | 2 months after surgery
  Determined with a validated IPSS questionnaire (in the corresponding language)
International Prostate Symptom Score (IPSS) | 1 year after surgery
  Determined with a validated IPSS questionnaire (in the corresponding language)
Quality of life | 2 months after surgery
  Determined with a validated QoL questionnaire (in the corresponding language)
Quality of life | 1 year after surgery
  Determined with a validated QoL questionnaire (in the corresponding language)
Maximal flow rate (Qmax) | 2 months after surgery
  Determined using uroflowmetry (ml/s)
Maximal flow rate (Qmax) | 1 year after surgery
  Determined using uroflowmetry (ml/s)
Voided volume (VV) | 2 months after surgery
  Determined using uroflowmetry (ml)
Voided volume (VV) | 1 year after surgery
  Determined using uroflowmetry (ml)
Catheter - free rate | 2 months after surgery
  Is the patient still having an indwelling or suprapubic catheter?
Catheter - free rate | 1 year after surgery
  Is the patient still having an indwelling or suprapubic catheter?

REFERENCES:
- [Background] Herrmann TR. Enucleation is enucleation is enucleation is enucleation. World J Urol. 2016 Oct;34(10):1353-5. doi: 10.1007/s00345-016-1922-3. Epub 2016 Sep 1. PMID 27585786
- [Background] Herrmann TR, Bach T, Imkamp F, Georgiou A, Burchardt M, Oelke M, Gross AJ. Thulium laser enucleation of the prostate (ThuLEP): transurethral anatomical prostatectomy with laser support. Introduction of a novel technique for the treatment of benign prostatic obstruction. World J Urol. 2010 Feb;28(1):45-51. doi: 10.1007/s00345-009-0503-0. PMID 20063164
- [Background] Herrmann TRW, Wolters M. Transurethral anatomical enucleation of the prostate with Tm:YAG support (ThuLEP): Evolution and variations of the technique. The inventors' perspective. Andrologia. 2020 Sep;52(8):e13587. doi: 10.1111/and.13587. Epub 2020 Apr 14. PMID 32286719
- [Background] Miernik A, Roehrborn CG. Benign Prostatic Hyperplasia Treatment On Its Way to Precision Medicine: Dream or Reality? Eur Urol Focus. 2022 Mar;8(2):363-364. doi: 10.1016/j.euf.2022.03.023. Epub 2022 Apr 7. No abstract available. PMID 35400612
- [Background] Gomez-Sancha F. The constant search for the greater good: evolving from TURP to anatomic enucleation of the prostate is a safe bet. World J Urol. 2021 Jul;39(7):2401-2406. doi: 10.1007/s00345-021-03637-1. Epub 2021 Feb 24. PMID 33625568
- [Background] Mitchell CR, Mynderse LA, Lightner DJ, Husmann DA, Krambeck AE. Efficacy of holmium laser enucleation of the prostate in patients with non-neurogenic impaired bladder contractility: results of a prospective trial. Urology. 2014 Feb;83(2):428-32. doi: 10.1016/j.urology.2013.09.035. Epub 2013 Nov 12. PMID 24231217
- [Background] Cho MC, Yoo S, Park J, Cho SY, Son H, Oh SJ, Paick JS. Effect of preoperative detrusor underactivity on long-term surgical outcomes of photovaporization and holmium laser enucleation in men with benign prostatic hyperplasia: a lesson from 5-year serial follow-up data. BJU Int. 2019 May;123(5A):E34-E42. doi: 10.1111/bju.14661. Epub 2019 Jan 27. PMID 30582661
- [Background] Aho T, Finch W, Jefferson P, Suraparaju L, Georgiades F. HoLEP for acute and non-neurogenic chronic urinary retention: how effective is it? World J Urol. 2021 Jul;39(7):2355-2361. doi: 10.1007/s00345-021-03657-x. Epub 2021 Mar 24. PMID 33763730